CLINICAL TRIAL: NCT00741728
Title: Heart Rate, Baroreflex Sensitivity and Cardiovascular Morbidity and Mortality in the Population. The Paris Prospective Study III
Brief Title: Heart Rate, Baroreflex Sensitivity and Cardiovascular Morbidity and Mortality in the Population
Acronym: PPSIII
Status: Active, not recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C07-39; 2007-A01386-47 (Registry Identifier: IDRCB)
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Community Based Study; Cardiovascular Disease; Sudden Death; Blood Pressure
Keywords: epidemiology; risk factors; heart rate; baroreflex sensitivity; sudden death
MeSH Terms: conditions — Cardiovascular Diseases; Death, Sudden | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and DNA taken from fresh blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- general population: Observational study of 10157 adult men and women from the general population who benefited from a free extensive health check up in Paris, France
  Interventions: Other: Spider flash ECG, high-precision carotid echo-tracking, step test

INTERVENTIONS:
Other: Spider flash ECG, high-precision carotid echo-tracking, step test — cardiac rhythm recorded during health check up, vascular aging parameters and baroreflex sensitivity recorded during carotid echotracking of the right common carotid artery , step test during 2 minutes

SUMMARY:
The aim of the present Paris Prospective Study III (PPS3) is (1) to assess the determinants of the regulation of heart rate and blood pressure variations and carotid properties (under different physiologic stimulations) and (2) to evaluate the respective contribution of heart rate, blood pressure variations and carotid properties to cardiovascular morbidity and mortality including sudden death during 10 years at least in healthy considered subjects.

DETAILED DESCRIPTION:
Overall, 10 157 men and women have been recruited during May 2008 and June 2012 for an extensive clinical examination including a 2h holter electrocardiography (ECG), a carotid doppler echo tracking, a step test, as well as blood and DNA collections. Since then, the cardiovascular morbidity and mortality of the participants is being followed up for 10 years at least and will continue up to 2032.

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years, French speaking, given consent for genetic analysis,
* written consent for participating in the study

Exclusion Criteria:

* <50 years and >75 years,
* no French speaking,
* current pregnancy,
* chronic severe disease,
* disagreement for genetic analysis,
* step test considered as non possible or non advisable by medical decision.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men and women affiliated to the public French Health Insurance System who benefited from a free general health check up paid by the French Health Insurance System
Sampling Method: Non-Probability Sample
Enrollment: 10157 (Actual)
Dates: Start 2008-05-13 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
cardiovascular disease (CVD) | through study completion, an average of 24 years
  incident coronary heart disease (CHD), stroke, sudden death, mortality

SECONDARY OUTCOMES:
heart rate parameters and baroreflex sensitivity | 4 Years
  as measured on the Spider Flash ECG and the carotid echotracking
other CVD outcomes | through study completion, an average of 24 years
  heart failure, arterial aneurysms, venous thromboembolism (VTE), pulmonary embolism, arrhythmic events (atrial fibrillation, flutter)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Jouven, MD, PhD, Study Director — INSERM and APHP; Jean-Philippe Empana, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Pierre Boutouyrie, MD, PhD, Principal Investigator — INSERM and APHP
Locations (1):
- Investigations Pré cliniques et Preventives de Paris, Paris, France

REFERENCES:
- [Background] Jouven X, Empana JP, Schwartz PJ, Desnos M, Courbon D, Ducimetiere P. Heart-rate profile during exercise as a predictor of sudden death. N Engl J Med. 2005 May 12;352(19):1951-8. doi: 10.1056/NEJMoa043012. PMID 15888695
- [Background] Jouven X, Zureik M, Desnos M, Courbon D, Ducimetiere P. Long-term outcome in asymptomatic men with exercise-induced premature ventricular depolarizations. N Engl J Med. 2000 Sep 21;343(12):826-33. doi: 10.1056/NEJM200009213431201. PMID 10995861
- [Background] Briet M, Bozec E, Laurent S, Fassot C, London GM, Jacquot C, Froissart M, Houillier P, Boutouyrie P. Arterial stiffness and enlargement in mild-to-moderate chronic kidney disease. Kidney Int. 2006 Jan;69(2):350-7. doi: 10.1038/sj.ki.5000047. PMID 16408126
- [Background] Kornet L, Hoeks AP, Janssen BJ, Houben AJ, De Leeuw PW, Reneman RS. Neural activity of the cardiac baroreflex decreases with age in normotensive and hypertensive subjects. J Hypertens. 2005 Apr;23(4):815-23. doi: 10.1097/01.hjh.0000163151.50825.e2. PMID 15775787
- [Background] Empana JP, Sykes DH, Luc G, Juhan-Vague I, Arveiler D, Ferrieres J, Amouyel P, Bingham A, Montaye M, Ruidavets JB, Haas B, Evans A, Jouven X, Ducimetiere P; PRIME Study Group. Contributions of depressive mood and circulating inflammatory markers to coronary heart disease in healthy European men: the Prospective Epidemiological Study of Myocardial Infarction (PRIME). Circulation. 2005 May 10;111(18):2299-305. doi: 10.1161/01.CIR.0000164203.54111.AE. Epub 2005 May 2. PMID 15867179
- [Derived] Alanis GA, Boutouyrie P, Abouqateb M, Bruno RM, Andrieu M, Vedie B, Geromin D, Danchin N, Laurent S, Jouven X, Empana JP. Accelerated Vascular Aging as a Possible Mechanism of Troponin I Release in the Absence of Clinically Manifested Myocardial Injury. J Am Heart Assoc. 2025 Apr;14(7):e037718. doi: 10.1161/JAHA.124.037718. Epub 2025 Mar 27. PMID 40145294
- [Derived] Deraz O, Range H, Boutouyrie P, Chatzopoulou E, Asselin A, Guibout C, Van Sloten T, Bougouin W, Andrieu M, Vedie B, Thomas F, Danchin N, Jouven X, Bouchard P, Empana JP. Oral Condition and Incident Coronary Heart Disease: A Clustering Analysis. J Dent Res. 2022 May;101(5):526-533. doi: 10.1177/00220345211052507. Epub 2021 Dec 7. PMID 34875909
- [Derived] Lisan Q, Tafflet M, Charles MA, Thomas F, Boutouyrie P, Guibout C, Haba-Rubio J, Perier MC, Pannier B, Marques-Vidal P, Jouven X, Empana JP. Self-reported body silhouette trajectories across the lifespan and excessive daytime sleepiness in adulthood: a retrospective analysis. The Paris Prospective Study III. BMJ Open. 2018 Mar 27;8(3):e020851. doi: 10.1136/bmjopen-2017-020851. PMID 29593025
- [Derived] Simon M, Boutouyrie P, Narayanan K, Gaye B, Tafflet M, Thomas F, Guibout C, Perier MC, Pannier B, Jouven X, Empana JP. Sex disparities in ideal cardiovascular health. Heart. 2017 Oct;103(20):1595-1601. doi: 10.1136/heartjnl-2017-311311. Epub 2017 Jul 28. PMID 28754808
- [Derived] Empana JP, Perier MC, Singh-Manoux A, Gaye B, Thomas F, Prugger C, Plichart M, Wiernik E, Guibout C, Lemogne C, Pannier B, Boutouyrie P, Jouven X. Cross-sectional analysis of deprivation and ideal cardiovascular health in the Paris Prospective Study 3. Heart. 2016 Dec 1;102(23):1890-1897. doi: 10.1136/heartjnl-2016-309502. Epub 2016 Jun 27. PMID 27354274
- See also: official website of the French National Institute for Health and Medical Research — http://www.inserm.fr